CLINICAL TRIAL: NCT03464617
Title: Doppler Flow Classification of Saint-Bonnet : A Non Interventional Clinical Trial
Brief Title: Doppler Flow Classification of Saint-Bonnet
Acronym: Saint-Bonnet
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_3099_SaintBonnet
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational Study that evaluates the interest of Doppler waveforms classification in Peripheral Artery disease

DETAILED DESCRIPTION:
Patients who have Doppler ultrasound scanning in clinical practice currently have a systematic record of Doppler flow on arterial axes of the aorta and right and left lower limbs. The investigators will analyze a posteriori Doppler flow of patients by classifying them using the 3 classifications. The patient will have no constraints related to this study since the recordings are currently performed in clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years;
* Social insured
* Patients referred in the department for any arterial examination of the lower limbs.

Exclusion Criteria:

- Patient unfit to understand the instructions of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients addressed in a vascular center for vascular ultrasound
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Doppler flows | Baseline
  The difference between the number of unclassified Doppler flows using the Saint-Bonnet classification and the number of unclassified flows using the Spronk et al. This comparison will be done using the Mc Nemar test.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU Amiens, Amiens
  - CHU de Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHU de Caen, Caen
  - CHU de Grenoble, Grenoble
  - CHU de Limoges, Limoges
  - CHU de Rennes, Rennes
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU de Toulouse, Toulouse
  - CH de Vichy, Vichy

IPD SHARING:
Plan to Share IPD: No